CLINICAL TRIAL: NCT07265102
Title: A Randomized Double-Blind Crossover Clinical Trial Evaluating the Efficacy of a Mouthwash Containing Chlorhexidine and Chlorine Dioxide in Patients With Oral Malodor
Brief Title: Effect of a Mouthwash Containing Chlorhexidine and Chlorine Dioxide on Halitosis
Acronym: CHX+CDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHXCDO-Halitosis-2022
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Halitosis
Keywords: halitosis; chlorhexidine; chlorine dioxide; mouthwash; volatile sulfur compounds; tongue coating
MeSH Terms: conditions — Halitosis | interventions — Cysteine Dioxygenase; Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both mouthwashes were packaged in identical opaque bottles labeled only with numerical codes (1 or 2) by an independent technician who was not involved in data collection or analysis. The two formulations were identical in appearance, color, odor, and taste to maintain blinding. The allocation code was kept confidential and sealed in an envelope until all data had been collected and statistical analyses were completed.
  Participants, clinicians, and outcome assessors were blinded to group allocation throughout the trial. Unblinding occurred only after all data analyses were completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHX-CDO Mouthwash (Experimental): Participants rinsed with a test mouthwash containing 0.01% chlorhexidine and 0.05% chlorine dioxide. Each participant used 15 mL of the solution twice daily (morning and evening) for 30 seconds over a period of 2 weeks. The mouthwash bottles were identical in appearance to maintain blinding.
  Interventions: Other: CHX 0.01% + CDO 0.05% mouthwash
- Placebo Mouthwash (Placebo Comparator): Participants rinsed with a placebo mouthwash containing the same excipients, color, and flavoring agents but without chlorhexidine or chlorine dioxide. Each participant used 15 mL of the placebo solution twice daily for 30 seconds over 2 weeks.
  Interventions: Other: Placebo mouthwash

INTERVENTIONS:
Other: CHX 0.01% + CDO 0.05% mouthwash — Mouthwash formulation containing chlorhexidine 0.01% and chlorine dioxide 0.05%, prepared by the Department of Pharmacy, University of Medicine and Pharmacy at Ho Chi Minh City.
  Other Names: CHX+ CDO mouthwash
  Arms: CHX-CDO Mouthwash
Other: Placebo mouthwash — Identical placebo formulation matched in flavor, color, and excipients but without active ingredients (CHX or CDO).
  Other Names: Control mouthwash
  Arms: Placebo Mouthwash

SUMMARY:
Halitosis significantly impacts the quality of a patient's life. This randomized, double-blind crossover trial evaluates a mouthwash containing chlorhexidine (0.01%) and chlorine dioxide (0.05%) compared with placebo. Forty participants rinsed twice daily for 2 weeks, followed by a 2-week washout and crossover. The primary outcomes were volatile sulfur compounds (H₂S, CH₃SH), measured by OralChroma. Secondary outcomes included plaque index, gingival index, bleeding on probing, tongue coating, and salivary bacterial counts (Aa, Pg, Fn, Pi, and Ec).

ELIGIBILITY:
Inclusion Criteria:

* ≥20 natural teeth
* H₂S >1.5 ng/10ml or CH₃SH >0.5 ng/10ml
* Signed informed consent

Exclusion Criteria:

* Systemic disease
* Smoking
* Pregnancy or lactation
* Periodontal pockets ≥4 mm
* Recent antibiotic use (<1 month)
* Orthodontic appliances or dentures
* Allergy to CHX or C

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Change in Hydrogen sulfide (H₂S) concentration in breath | baseline, immediate post-rinse, 2 weeks
  The concentration of hydrogen sulfide (H₂S) in oral breath was measured using the OralChroma™ device. The difference between baseline, immediately after rinsing, and 2 weeks was used to assess the efficacy of the mouthwash in reducing volatile sulfur compounds.
Change in Methyl mercaptan (CH₃SH) concentration in breath | Baseline, immediate post-rinse, 2 weeks
  The concentration of methyl mercaptan (CH₃SH) in oral breath was measured using the OralChroma™ device. The difference between baseline, immediately after rinsing, and 2 weeks was used to evaluate the short-term and sustained effects of the mouthwash on halitosis.

SECONDARY OUTCOMES:
Change of plaque index | At baseline and 2 weeks of mouthwash use
  The Plaque Index (PI) was recorded at four surfaces per tooth (mesiobuccal, buccal, distobuccal, and lingual) to assess plaque accumulation. Each surface was scored on a scale from 0 to 3, where 0 indicates no plaque and 3 indicates abundant plaque accumulation. The mean PI score per participant was calculated at each visit. A lower score indicates less plaque accumulation and improved oral hygiene.
Change in Gingival Index (GI) | At baseline and 2 weeks of mouthwash use
  The Gingival Index (GI) was evaluated at four surfaces per tooth (mesiobuccal, buccal, distobuccal, and lingual) to assess the degree of gingival inflammation. Each surface was scored on a scale from 0 to 3, where 0 indicates normal gingiva and 3 indicates severe inflammation with marked redness, edema, and a tendency to spontaneous bleeding. The mean GI score per participant was calculated. A lower score reflects healthier gingival conditions.
Change in Bleeding on Probing (BOP) | At baseline and 2 weeks of mouthwash use
  The percentage of sites showing bleeding upon gentle probing was recorded as an indicator of gingival inflammation and bleeding tendency. The presence of bleeding was recorded at each examined site following gentle periodontal probing. BOP was expressed as the percentage of bleeding sites, calculated as the number of sites showing bleeding divided by the total number of sites examined ×100%. Higher percentages indicate greater gingival inflammation.
Change in Tongue Coating Index | At baseline and 2 weeks of mouthwash use
  The tongue dorsum was visually divided into six areas (three anterior and three posterior) according to Winkel's Tongue Coating Index (WTCI). Each area was scored from 0 (no coating), 1 (mild coating), and 2 (thick coating), and the total score (0-12) was calculated as the Tongue Coating Index.
Change in salivary bacterial load (qPCR quantification) | At baseline and 2 weeks of mouthwash use
  Salivary bacterial counts of Porphyromonas gingivalis, Fusobacterium nucleatum, Prevotella intermedia, Eikenella corrodens, and Aggregatibacter actinomycetemcomitans were quantified using real-time PCR (qPCR). Changes in bacterial load (log CFU/mL) between baseline and 2 weeks were compared to assess the antibacterial effect of the mouthwash.

CONTACTS AND LOCATIONS:
Overall Officials: Thuy A.V. Pham, Assoc.Prof., Principal Investigator — Can Tho University of Medicine and Pharmacy
Locations (1):
- Odonto-Stomatology Hospital of Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
De-identified data, study protocol, and statistical code will be available upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: Within 6 months after publication, available for 3 years
Access Criteria: Researchers with IRB-approved proposals may request access via corresponding author.

REFERENCES:
- [Background] Pham TAV, Nguyen NTX. Efficacy of chlorine dioxide mouthwash in reducing oral malodor: A 2-week randomized, double-blind, crossover study. Clin Exp Dent Res. 2018 Oct 23;4(5):206-215. doi: 10.1002/cre2.131. eCollection 2018 Oct. PMID 30386642
- [Background] Shinada K, Ueno M, Konishi C, Takehara S, Yokoyama S, Zaitsu T, Ohnuki M, Wright FA, Kawaguchi Y. Effects of a mouthwash with chlorine dioxide on oral malodor and salivary bacteria: a randomized placebo-controlled 7-day trial. Trials. 2010 Feb 12;11:14. doi: 10.1186/1745-6215-11-14. PMID 20152022